CLINICAL TRIAL: NCT05601960
Title: A Combination of a Dermocosmetic and a Tainted Sunscreen Reduce Acne Severity and Signs of Post-inflammatory Hyperpigmentation in Subjects With a Fitzpatrick Phototype Ranging From IV to VI
Brief Title: A Combination Treatment Reduces Acne Severity and PIHP
Status: Completed | Type: Observational
Sponsor: Cosmetique Active International (Industry)
Responsible Party: Sponsor
Other Study IDs: LRP19009
Record Dates: First submitted 2022-10-25; First posted 2022-11-01 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Acne; Postinflammatory Hyperpigmentation
MeSH Terms: conditions — Acne Vulgaris; Hyperpigmentation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: anti-acne dermocosmetic — Topical application once daily for 2 months
  Other Names: Sun screen

SUMMARY:
Acne is a chronic, inflammatory skin condition. It may cause scars and post-inflammatory hyperpigmentation (PIHP). PIHP frequently affects individuals with a phototype of IV or above.[1] PIHP is worsened by UV radiation, lasts for years and impacts the individual well-being.[2, 3] In an observational study, 1785 adults with a phototype ranging from IV to VI with acne and PIHP applied daily for 2 months a dermocosmetic and a tainted sunscreen product (DC, Effaclar® Duo (+); SS, Anthelios® Shaka Fluide SPF 50+, SS; both La Roche-Posay Laboratoire Dermatologique, France.

ELIGIBILITY:
Inclusion Criteria:

* adult
* mild to moderate acne
* presence of postinflammatory hyperpigmentation lesions
* phototype IV to VI

Exclusion Criteria:

* less than 18 years
* severe acne

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult subjects with mild to moderate acne, post-inflammatory hyperpigmentation and of any phototype were suitable for this study.
Sampling Method: Non-Probability Sample
Enrollment: 1785 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
seborrhoea level | baseline
  visual analog scale scale 0=none to 10= very severe
seborrhoea level | Month 2
  visual analog scale 0=none to 10= very severe
acne severity | baseline
  GEA (Global evaluation of acne) scale 0=none to 5=very severe
acne severity | Month 2
  GEA (Global evaluation of acne) scale 0=none to 5=very severe
PAHPI: post-acne hyperpigmentation index | baseline
  post-acne hyperpigmentation index from <3mm to >10mm
PAHPI: post-acne hyperpigmentation index | Month 2
  post-acne hyperpigmentation index from <3mm to >10mm
inflammatory lesions | baseline
  lesion count
inflammatory lesions | Month 2
  lesion count
non-inflammatory lesions | baseline
  lesion count
non-inflammatory lesions | Month 2
  lesion count

SECONDARY OUTCOMES:
Investigator satisfaction acne | Month 2
  visual analog scale from very unsatified=0 to very satisfied=5
Investigator satisfaction | Month 2
  visual analog scale from very unsatified=0 to very satisfied=5
Patient satisfaction acne | Month 2
  visual analog scale from very unsatified=0 to very satisfied=5
Patient satisfaction PAHPI | Month 2
  visual analog scale from very unsatified=0 to very satisfied=5
Patient: Skin quality | Month 2
  visual analog scale from very unsatified=0 to very satisfied=5

CONTACTS AND LOCATIONS:
Overall Officials: Rana Shabab, Principal Investigator — Dermatique Skin Care, Khobar, KSA
Locations (1):
- L'Oreal, Dubai, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No